CLINICAL TRIAL: NCT00217997
Title: Impulsivity, Brain Function and Substance Abuse Treatment
Brief Title: Impulsivity, Brain Function, and Substance Abuse Treatment in Cocaine Dependent Individuals
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Texas (Other)
Responsible Party: Sponsor
Other Study IDs: NIDA-09262-6; 5P50DA009262-17 (NIH); P50-09262-6; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Cocaine Abuse; Cocaine-Related Disorders
Keywords: cocaine abuse; Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cocaine dependence is a major public health problem; an effective primary treatment for cocaine dependent individuals has yet to be found. The purpose of this trial is to evaluate aspects of treatment response in cocaine dependent individuals.

DETAILED DESCRIPTION:
Cocaine is a strong central nervous system stimulant that is widely abused throughout the United States. Due to its widespread use, it is important to develop an effective treatment for cocaine dependence. The purpose of this study is to determine how impulsivity and prefrontal cortical function are related to treatment response in cocaine dependent individuals.

Participants in this study will complete four separate experiments, each with a different aim and testing panel [cognitive function tests with and without functional magnetic resonance imaging (fMRI)]. The first experiment will examine memory, attention, cognitive function, and impulsivity; the aim is to determine the relationship between impulsivity and cognitive function in cocaine dependent individuals receiving treatment. The second experiment will examine the relationship between impulsivity and the prefrontal cortical structure and function. Participants will complete an fMRI during the second experiment. The third experiment will consist of cognitive function tests and will examine the prefrontal cortex in relation to treatment response, based on four different treatments: 1) L-dopamine, 2) naltrexone, 3) modafinil, and 4) placebo. The fourth experiment will examine the effect of cocaine dependence treatment on prefrontal cortex, focusing on participants receiving modafinil.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for cocaine dependence
* Met inclusion criteria for other cocaine dependence studies within the center grant

Exclusion Criteria:

* Current or history of DSM-IV Axis I disorders, other than substance abuse or dependence
* Lifetime diagnosis of alcohol dependence
* Serious non-psychiatric medical illness requiring ongoing medical treatment or one that affects the central nervous system
* Positive urine drug screen test for drugs of abuse other than cocaine at the time of study entry
* AIDS-defining illness
* Intelligence Quotient (IQ) below 70
* Pregnant
* Uses a pacemaker, metal or electromechanical implants, or metallic foreign bodies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cocaine Dependent Subjects
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2005-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
fMRI brain activation | baseline
  Baseline predictor of treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Frederick G. Moeller, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States

REFERENCES:
- [Background] Orru M, Guitart X, Karcz-Kubicha M, Solinas M, Justinova Z, Barodia SK, Zanoveli J, Cortes A, Lluis C, Casado V, Moeller FG, Ferre S. Psychostimulant pharmacological profile of paraxanthine, the main metabolite of caffeine in humans. Neuropharmacology. 2013 Apr;67:476-84. doi: 10.1016/j.neuropharm.2012.11.029. Epub 2012 Dec 19. PMID 23261866
- [Background] Liu S, Lane SD, Schmitz JM, Green CE, Cunningham KA, Moeller FG. Increased intra-individual reaction time variability in cocaine-dependent subjects: role of cocaine-related cues. Addict Behav. 2012 Feb;37(2):193-7. doi: 10.1016/j.addbeh.2011.10.003. Epub 2011 Oct 12. PMID 22047976
- [Background] Ma L, Steinberg JL, Hasan KM, Narayana PA, Kramer LA, Moeller FG. Working memory load modulation of parieto-frontal connections: evidence from dynamic causal modeling. Hum Brain Mapp. 2012 Aug;33(8):1850-67. doi: 10.1002/hbm.21329. Epub 2011 Jun 20. PMID 21692148
- [Background] Liu S, Lane SD, Schmitz JM, Waters AJ, Cunningham KA, Moeller FG. Relationship between attentional bias to cocaine-related stimuli and impulsivity in cocaine-dependent subjects. Am J Drug Alcohol Abuse. 2011 Mar;37(2):117-22. doi: 10.3109/00952990.2010.543204. Epub 2011 Jan 5. PMID 21204739
- [Background] Lane SD, Steinberg JL, Ma L, Hasan KM, Kramer LA, Zuniga EA, Narayana PA, Moeller FG. Diffusion tensor imaging and decision making in cocaine dependence. PLoS One. 2010 Jul 16;5(7):e11591. doi: 10.1371/journal.pone.0011591. PMID 20661285
- [Background] Narayana PA, Datta S, Tao G, Steinberg JL, Moeller FG. Effect of cocaine on structural changes in brain: MRI volumetry using tensor-based morphometry. Drug Alcohol Depend. 2010 Oct 1;111(3):191-9. doi: 10.1016/j.drugalcdep.2010.04.012. Epub 2010 May 31. PMID 20570057
- [Background] Schmitz JM, Mooney ME, Green CE, Lane SD, Steinberg JL, Swann AC, Moeller FG. Baseline neurocognitive profiles differentiate abstainers and non-abstainers in a cocaine clinical trial. J Addict Dis. 2009 Jul;28(3):250-7. doi: 10.1080/10550880903028502. PMID 20155594